CLINICAL TRIAL: NCT06385665
Title: The Effect of Appropriate Family Companionship on the Physical and Mental Health of Patients With Advanced Breast Cancer:A Real World Study
Brief Title: The Effect of Appropriate Family Companionship on the Physical and Mental Health of Patients With Advanced Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin Peng (Other)
Responsible Party: Sponsor-Investigator, Xin Peng, Deputy chief nurse, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Xin Peng
Record Dates: First submitted 2023-12-26; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accompanying group (Experimental)
  Interventions: Behavioral: Graded companionship
- non-accompanied group (No Intervention)

INTERVENTIONS:
Behavioral: Graded companionship — Accompanying levels are divided into beginner, intermediate and advanced
  Arms: accompanying group

SUMMARY:
The goal of this clinical trial is to learn about companionship needs in breast cancer patients who are pathologically or cytologically diagnosed as cancer, are alive with the tumor, and have TNM clinical stage IV. The main questions it aims to answer are:

1. Patients with advanced breast cancer need family companionship
2. Analyze and study the reasons and factors that affect the physical and mental impact of effective family companionship on patients with advanced breast cancer Participants will be divided into a companion group and a non-accompaniment group. Patients in the companion group are given graded companion intervention methods. A comparison group: Researchers will compare a non-accompaniment group to see if the physical and mental impact of companionship on patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who are pathologically or cytologically diagnosed as cancer
* TNM clinical stage IV

Exclusion Criteria:

* Terminal cancer patients who are mentally ill or confused and refuse to participate in the survey

Ages: 21 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline meatal state on GAD-7 at Week 48. | Baseline and Week 48
  The GAD-7 is a validated, self-reported instrument assessing average mental state intensify over the past 24 hour period. Possible scores range from 0 to 21.Change = (Week 48 Score - Baseline Score)
Change from Baseline physical state on kps at Week 48. | Baseline and Week 48
  The kps is a validated, self-reported instrument assessing physical state average intensify over the past 24 hour period. Possible scores range from 0 to 100.Change = (Week 48 Score - Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Deyin Hu, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes